CLINICAL TRIAL: NCT05151133
Title: Clinical Study of Moderate to Severe Persistent Allergic Rhinitis Therapy by Human Umbilical Cord Mesenchymal Stem Cells
Brief Title: Clinical Study of Allergic Rhinitis Therapy by Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-002
Record Dates: First submitted 2021-11-10; First posted 2021-12-09 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Allergic Rhinitis
Keywords: Umbilical cord; Mesenchymal Stem Cells; Allergic Rhinitis; Therapy
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose UCMSCs (Experimental)
  Interventions: Biological: Low dose UCMSCs
- Moderate dose UCMSCs (Experimental)
  Interventions: Biological: Moderate dose UCMSCs
- High dose UCMSCs (Experimental)
  Interventions: Biological: High dose UCMSCs

INTERVENTIONS:
Biological: Low dose UCMSCs — Receive one course of treatment with a single injection : 0.5×10^6 cells/kg, with a total volume of 100 ml UCMSCs;
  Arms: Low dose UCMSCs
Biological: Moderate dose UCMSCs — Receive one course of treatment with a single injection : 1.0×10^6 cells/kg, with a total volume of 100 ml UCMSCs;
  Arms: Moderate dose UCMSCs
Biological: High dose UCMSCs — Receive one course of treatment with a single injection : 2.0×10^6 cells/kg, with a total volume of 100 ml UCMSCs;
  Arms: High dose UCMSCs

SUMMARY:
The investigators is now carrying out a clinical study of Umbilical cord Mesenchymal Stem Cells (UCMSCs) in the treatment of Allergic rhinitis (AR). UCMSCs is known to its multilineage differentiation potential, strong proliferation ability, low immunogenicity, convenient material acquisition, and fewer restrictions on ethical and moral issues. The investigators hope to find a novel, minimally invasive, effective and simple treatment for the large number of patients with persistent moderate to severe AR.

DETAILED DESCRIPTION:
Allergic rhinitis (AR), is a noninfectious inflammatory disease of nasal mucosa mediated by immunoglobulin E (IgE) antibody and involved in a variety of immune active cells and cytokines after the atopic body is exposed to allergens. The incidence of allergic rhinitis increases as people's living standards improves. It is estimated that about 1.4 billion people worldwide have been affected by the disease. Some patients with moderate to severe AR have no improvement in symptoms after drug treatment, which continues to affect daily life and work. Therefore, these patients urgently needs a new, minimally invasive, effective and simple treatment. Mesenchymal Stem Cells (MSCs) are pluripotent stem cells derived from the mesoderm, which can differentiate into bone, cartilage, fat and other cells. MSCs can also secrete a variety of bioactive molecules, which have the effects of regulating immunity and anti-inflammatory. Based on its immunomodulatory effect, MSCs is gradually becoming a new star in the treatment of allergic diseases. In pre-clinical studies on the treatment of AR, MSCs have shown good therapeutic effect in the treatment of allergic rhinitis.

This study is a prospective, open, single-center clinical study. Participants were recruited into three different dose groups. The cohort size of each dose group was 6 participants. The subjects of each group each will receive one course of treatment with a single injection. Subjects of group 1 will receive 0.5×10^6 cells/kg, with a total volume of 100 ml UCMSCs; group 2 will receive 1.0×10^6 cells/kg; with a total volume of 100 ml UCMSCs; group 3 will receive 2.0×10^6 cells/kg, with a total volume of 100 ml UCMSCs. One month after each injection, the Data and Safety Monitoring Committee (DSMC) will comprehensively evaluate the results of the phased clinical research, and after determining the safety and feasibility of the research, the enrollment of the next phase will start. The subjects will be followed up on the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment. The main outcome measures are the severity and incidence of adverse events. The secondary outcome measures are RQLQ score, VAS score, serum inflammatory factor detection, nasal secretion inflammatory factor detection, nasal function test and nasal endoscopy, etc. In addition, the investigators will also monitor safety indicators such as blood routine, urine routine, liver and kidney function, immunological indicators, tumor markers, etc. At the end of the study, according to the data obtained, the clinical safety and feasibility of intravenous infusion of UCMSCs in the treatment of moderate to severe persistent AR will be evaluated, so as to provide drug dose basis for the next stage of clinical research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with moderate to severe persistent allergic rhinitis who meet the diagnostic criteria for allergic rhinitis (2015 Tianjin standard);
2. The results of allergen examination showed that the allergen was a single allergy of dust mite;
3. After more than 2 years of antihistamine, nasal glucocorticoid and other drug treatments, the curative effect is poor, and the symptoms seriously affect the patient's life;
4. Age 18-60 years old;
5. The patient refused to receive allergen-specific immunotherapy;
6. The patient is willing to receive stem cell therapy and sign an informed consent.

Exclusion Criteria:

1. The subject is accompanied by sinusitis, asthma and aspirin intolerance;
2. The subjects suffer from severe primary heart, liver, lung, kidney and blood diseases;
3. The subjects suffer from Malignant tumors;
4. The subjects suffer from severe immune diseases;
5. The subjects suffer from mental illness;
6. Female subjects who are or are about to become pregnant, pregnant or breastfeeding;
7. Patients who are participating in other clinical trials;
8. In addition to the above conditions, there are other reasons why researchers believe that they are not suitable to participate in this clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Severity and incidence of adverse events (SIAE) on the day of treatment | Day 1 of treatment
  The assessment was conducted according to the Common Adverse Event Evaluation Standard 4.0 (NCI-CTCAE v4.0) jointly issued by the U.S. Department of Health and Human Services, the National Institutes of Health, and the National Cancer Institute.
3rd day SIAE | 3 days after treatment
  The assessment was conducted according to the Common Adverse Event Evaluation Standard 4.0 (NCI-CTCAE v4.0) jointly issued by the U.S. Department of Health and Human Services, the National Institutes of Health, and the National Cancer Institute.
1 week SIAE | 1 week after treatment
  The assessment was conducted according to the Common Adverse Event Evaluation Standard 4.0 (NCI-CTCAE v4.0) jointly issued by the U.S. Department of Health and Human Services, the National Institutes of Health, and the National Cancer Institute.
1 month SIAE | 1 month after treatment
  The assessment was conducted according to the Common Adverse Event Evaluation Standard 4.0 (NCI-CTCAE v4.0) jointly issued by the U.S. Department of Health and Human Services, the National Institutes of Health, and the National Cancer Institute.
3 months SIAE | 3 months after treatment
  The assessment was conducted according to the Common Adverse Event Evaluation Standard 4.0 (NCI-CTCAE v4.0) jointly issued by the U.S. Department of Health and Human Services, the National Institutes of Health, and the National Cancer Institute.
6 months SIAE | 6 months after treatment
  The assessment was conducted according to the Common Adverse Event Evaluation Standard 4.0 (NCI-CTCAE v4.0) jointly issued by the U.S. Department of Health and Human Services, the National Institutes of Health, and the National Cancer Institute.
12 months SIAE | 12 months after treatment
  The assessment was conducted according to the Common Adverse Event Evaluation Standard 4.0 (NCI-CTCAE v4.0) jointly issued by the U.S. Department of Health and Human Services, the National Institutes of Health, and the National Cancer Institute.
24 months SIAE | 24 months after treatment
  The assessment was conducted according to the Common Adverse Event Evaluation Standard 4.0 (NCI-CTCAE v4.0) jointly issued by the U.S. Department of Health and Human Services, the National Institutes of Health, and the National Cancer Institute.

SECONDARY OUTCOMES:
RQLQ score | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  The assessment of Rhinoconjunctivitis quality of life questionnaire (RQLQ) includes daily activities, sleep, non-rhino-conjunctivitis symptoms, rhinitis-related behaviors, nasal symptoms, eye symptoms, and emotional reactions.
  Each of the above aspect is composed of several measurements. A total of 28 measurements are individually scored from 0 to 6 points. A score of 0 indicates that the subject has not been affected by nose and eye symptoms in the past week, a score of 1 indicates that it is almost unaffected, a score of 2 indicates a minor influence, a score of 3 indicates a slight influence, a score of 4 indicates a moderate influence, and a score of 5 indicates a severe influence, a score of 6 indicates that it is extremely severely affected. In terms of daily activities, a score of 9 directly indicates that daily activity cannot be carried out due to nose and eye symptoms.
VAS score | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  Visual analogue scale (VAS) is used to evaluate the severity of nasal symptoms by patients or their guardians. Visual line marks are made on the scale with a length of 10 cm. The VAS score is calculated as 0 is asymptomatic (0 cm), and 10 is the most serious symptom (10 cm).
Nasal function test | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  Nasal expiratory nitric oxide (NO) test (NNO test), is a simple, noninvasive and convenient medical detection method, that can be used for the diagnosis, treatment and monitoring of nasal diseases such as rhinitis, sinusitis and nasal polyps.
Nasal endoscopy | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  The normal nasal mucosa is light red, with smooth, moist and shiny surface. The nasal cavity and nasopharyngeal mucosa have no congestion, edema, dryness, ulcers, hemorrhage, vasodilatation and new organisms; no purulent secretions.
  The mucosa of allergic rhinitis is pale, edematous or lavender, and the discharge is watery.
U-HCG | The day of enrollment screening, 3 months, 6 months, 12 months, and 24 months after the treatment.
  The U-HCG test detects levels of hCG in the urine, positive result indicate pregnacy.
Detection of Serum Interferon γ (IFN-γ) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interferon γ (IFN-γ) in the serum;
Detection of Serum Interferon α (IFN-α) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interferon α (IFN-α) in the serum;
Detection of Serum Interleukin 1β (IL-1β) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 1β (IL-1β) in the serum;
Detection of Serum Interleukin 2 (IL-2) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 2 (IL-2) in the serum;
Detection of Serum Interleukin 4 (IL-4) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 4 (IL-4) in the serum;
Detection of Serum Interleukin 5 (IL-5) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 5 (IL-5) in the serum;
Detection of Serum Interleukin 6 (IL-6) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 6 (IL-6) in the serum;
Detection of Serum Interleukin 8 (IL-8) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 8 (IL-8) in the serum;
Detection of Serum Interleukin 10 (IL-10) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 10 (IL-10) in the serum;
Detection of Serum Interleukin 12P70 (IL-12P70) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 12P70 (IL-12P70) in the serum;
Detection of Serum Interleukin 17A (IL-17A) | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 17A (IL-17A) in the serum;
Detection of Serum Tumor necrosis factor-α（TNF-α） | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Tumor necrosis factor-α（TNF-α） in the serum;
Detection of inflammatory factor Interferon γ (IFN-γ) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interferon γ (IFN-γ) in nasal secretions;
Detection of inflammatory factor Interferon α (IFN-α) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interferon α (IFN-α) in nasal secretions;
Detection of inflammatory factor Interleukin 1β (IL-1β) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interferon α (IFN-α) in nasal secretions;
Detection of inflammatory factor Interleukin 2 (IL-2) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 2 (IL-2) in nasal secretions;
Detection of inflammatory factor Interleukin 4 (IL-4) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 4 (IL-4) in nasal secretions;
Detection of inflammatory factor Interleukin 5 (IL-5) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 5 (IL-5) in nasal secretions;
Detection of inflammatory factor Interleukin 6 (IL-6) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 6 (IL-6) in nasal secretions;
Detection of inflammatory factor Interleukin 8 (IL-8) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 8 (IL-8) in nasal secretions;
Detection of inflammatory factor Interleukin 10 (IL-10) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 10 (IL-10) in nasal secretions;
Detection of inflammatory factor Interleukin 12P70 (IL-12P70) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 12P70 (IL-12P70) in nasal secretions;
Detection of inflammatory factor Interleukin 17A (IL-17A) in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Interleukin 17A (IL-17A) in nasal secretions;
Detection of inflammatory factor Tumor necrosis factor-α（TNF-α） in nasal secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To test level of inflammatory factor Tumor necrosis factor-α（TNF-α） in nasal secretions;

OTHER OUTCOMES:
Blood routine | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  Include hemoglobin determination, red blood cell count, white blood cell count white blood cell classification.
Urine routine | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  Include urine color, potential of hydrogen (pH) value of urine, protein qualitative and microscopic determination of urine sediment count.
Liver and kidney function | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  A group of laboratory tests that helps detect problems or disorders in the liver or kidney.
Immunological indicators | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  Cell counts of T cells and their subtypes in peripheral blood
Tumor markers | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  Carcinoembryonic antigen（CEA） ，Alpha-FetoProtein（AFP）
Total Protein Concentration of Nasal Secretions | The day of enrollment screening, the 3rd day, 1 week, 1 month, 3 months, 6 months, 12 months, and 24 months after the treatment.
  To determinate the total protein concentration of nasal secretions.

CONTACTS AND LOCATIONS:
Overall Officials: Xicheng Song, MD, Principal Investigator — Yantai Yuhuangding Hospital
Locations (1):
- Yantai Yuhuangding Hospital, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: No